CLINICAL TRIAL: NCT00451282
Title: Stepped Preventive Care to Reduce the Impact of Acute Pediatric Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2006-9-4974; R49CE000987-01 (NIH)
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Results first posted 2015-04-20 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Stress Disorders, Posttraumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stepped Preventive Care (Experimental): Receiving Stepped Preventive Care intervention - at least 2 brief assessments with nurse and/or social worker (1) during hospital admission , and (2) approximately 2 weeks post-discharge. Additional interventions provided as needed, based on manual.
  Interventions: Behavioral: stepped preventive care
- Treatment as usual (No Intervention): Medical and psychosocial care per usual hospital protocols, which may include social work support.

INTERVENTIONS:
Behavioral: stepped preventive care — 2 targeted assessments (T1: in hospital within a few days of injury; T2: two weeks post-discharge) are administered by nurse or social worker, and determine need for additional assistance modules. Additional modules include case management, care coordination, assistance with child and family coping with injury/distress, and trauma-focused Cognitive Behavior Therapy (CBT) beginning at 4-6 weeks post-injury if needed.
  Arms: Stepped Preventive Care

SUMMARY:
This study will evaluate the impact of a brief psychosocial intervention delivered to children or adolescents who are hospitalized for an unintentional injury. The intervention is designed to promote psychological recovery and enhance functional outcomes after injury. The study will also provide preliminary data concerning cost-effectiveness of the intervention.

The core study hypotheses are that children receiving the intervention will (1) have lower severity of post-traumatic stress disorder (PTSD) and depression symptoms at follow-up; (2) show greater adherence to discharge instructions and better health-related quality of life at follow-up, and (3) have higher rates of attendance at scheduled follow-up appointments and lower rates of emergency room utilization and re-hospitalization in the 6 months post-injury, compared to those receiving usual care.

DETAILED DESCRIPTION:
The purpose of this study is to examine the effectiveness of a stepped care model for prevention of psychosocial distress (especially posttraumatic stress) after injury. The model includes screening for risk, standard follow-up with those at risk, and additional evidence-based interventions matched to individual need.

The study will evaluate the impact of the intervention on psychosocial outcomes (PTSD and depression symptoms); as well as health outcomes (adherence to discharge instructions, health-related quality of life), and will provide preliminary data to inform cost-effectiveness analyses by describing the costs of providing the intervention and examining its impact on subsequent health service utilization.

Study Design: 180 children at risk for persistent psychosocial distress post-injury, based on a screening assessment, will be randomized to the Stepped Preventive Care intervention or usual care. An additional comparison group of 90 low risk children will also receive usual care and be followed for assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age 8 to 17
* Admitted to hospital for treatment of unintentional injury
* Sufficient English fluency to participate in an interview
* Family has access to a telephone (for telephone follow-up contacts)

Exclusion criteria:

* Child's medical status or cognitive functioning precludes participating in an interview
* Child has moderate to severe head injury, defined as Glasgow Coma Score (GCS) <= 12
* Child's injury involved family violence or abuse (physical or sexual)
* No parent or guardian available to consent

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 290 (Actual)
Dates: Start 2007-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Kassam-Adams, PhD, Principal Investigator — Center for Injury Research and Prevention, Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Kassam-Adams N, Garcia-Espana JF, Marsac ML, Kohser KL, Baxt C, Nance M, Winston F. A pilot randomized controlled trial assessing secondary prevention of traumatic stress integrated into pediatric trauma care. J Trauma Stress. 2011 Jun;24(3):252-9. doi: 10.1002/jts.20640. Epub 2011 May 18. PMID 21594900

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potentially eligible injured patients were identified from patient census and administration lists (n=1330; April 2007 - October 2008). Of 845 eligible children, 149 refused participation, 406 were not approached, usually due to limited parent availability.
Pre-assignment Details: 290 children were enrolled for risk screening, of these 85 (29%) scored positive on one or more screening measures for PTSD and were randomly assigned to receive usual care or the intervention (n=39 and n=46 respectively). 5 intervention subjects did not end up receiving the allocated intervention.
Groups:
- Intervention: Injured children receiving Stepped Preventive Care intervention
- Usual Care: Injured children receiving usual care
Period: Overall Study
Arm/Group | Intervention | Usual Care
Started | 46 | 39
Completed | 40 | 34
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 46 | 39 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 46 | 39 | 85
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.2 (2.2) | 11.9 (2.7) | 11.5 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 11 | 34
  Male | 23 | 28 | 51
Region of Enrollment [Number; unit: participants]
  United States | 46 | 39 | 85

OUTCOME MEASURES:

1. Primary Outcome: PTSD Symptoms in Children 6 Weeks Post-injury
Description: The Child PTSD Symptom Scale (CPSS) is a 24-item self-report instrument that yields both a continuous severity score and a determination of likely PTSD diagnostic status according to symptom presence. 17 items corresponding to of the Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV symptom criteria (and are assumed to yield a PTSD symptom severity score range 0-51) and 7 items assess impairment from those symptoms. The 17 symptom items were administered at baseline (prerandomization), with a score of 15 or greater considered a positive screen for PTSD risk (higher values represent more significant severity of and impairment from PTSD symptoms). The 24-item scale was administered at 6 weeks and 6 months postinjury to assess traumatic stress symptom outcomes.
Time Frame: 6 weeks
Population: 85 children were randomly assigned to receive usual care (n=39) or the intervention (n=46, 5 did not go on to receive intervention). Of these subjects, 28 usual care subjects and 36 intervention subjects completed 6 week follow-up.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 36 | 28
Units on a scale | 12.6 (10.2) | 13.6 (10.7)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority or Other; p = .69, t-test, 2 sided

2. Primary Outcome: PTSD Symptoms in Children 6 Months Post-injury
Description: The Child PTSD Symptom Scale (CPSS) is a 24-item self-report instrument that yields both a continuous severity score and a determination of likely PTSD diagnostic status according to symptom presence. 17 items corresponding to DSM-IV symptom criteria (and are assumed to yield a PTSD symptom severity score range 0-51) and 7 items assess impairment from those symptoms. The 17 symptom items were administered at baseline (prerandomization), with a score of 15 or greater considered a positive screen for PTSD risk (higher values represent more significant severity of and impairment from PTSD symptoms). The 24-item scale was administered at 6 weeks and 6 months postinjury to assess traumatic stress symptom outcomes.
Time Frame: 6 months
Population: 85 children were randomly assigned to receive usual care (n=39) or the intervention (n=46, 5 did not go on to receive intervention). Of these subjects, 31 usual care subjects and 37 intervention subjects completed 6 month follow-up.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 37 | 31
Units on a scale | 12.6 (11.6) | 12.2 (9.7)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority or Other; p = .89, t-test, 2 sided

3. Secondary Outcome: Depression Symptoms in Children 6 Wks Post-injury
Description: The Center for Epidemiologic Studies Depression Scale (CES-D) is a 20-item self-report measure of depression symptoms that yields a total severity score (range 0-60) . Clinical cut-off scores (≥16 for adults and ≥24 for youth) have been empirically established. Higher values represent more significant severity of symptoms of depression. The CES-D has been validated in adults and children 10 and over as an effective screen for depression. The CES-D was administered at baseline (prerandomization), 6 weeks and 6 months postinjury.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 36 | 28
Units on a scale | 15.0 (10.7) | 14.0 (10.8)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority or Other; p = .69, t-test, 2 sided

4. Secondary Outcome: Depression Symptoms in Children 6 Mos Post-injury
Description: as for outcome 3
Time Frame: 6 months
Population: 85 children were randomly assigned to receive usual care (n=39) or the intervention (n=46, 5 did not go on to receive intervention). Of these subjects, 31 usual care subjects and 37 intervention subjects completed 6 week follow-up.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 37 | 31
Units on a scale | 15.6 (13.8) | 11.6 (9.9)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority or Other; p = .18, t-test, 2 sided

5. Secondary Outcome: Health-related Quality of Life 6 Weeks and 6 Months Post-injury
Description: The Pediatric Quality of Life Inventory is a well-validated measure of child health-related quality of life. Children completed the measure at baseline to report preinjury functioning and at 6-weeks and 6-months postinjury regarding current functioning. Current analyses utilize the 8-item Physical health/Physical functioning subscale. Scores range from 0-100; higher scores indicate better functioning outcomes.
Time Frame: 6 months
Reporting Status: Not Posted

6. Secondary Outcome: Adherence With Medical Discharge Instructions
Description: The Health Care Questionnaire for Parents, created for this study, will assess health services utilized post-injury, adherence with specific discharge instructions (e.g., attendance at recommended follow-up appointments), as well as the number of days missed from work (parent) or school (child) related to the injury. Outcome variables to assess adherence will be dichotomized (e.g., attended scheduled appt? yes / no). The Health Care Questionnaire for Primary Care Physicians (PCPs) will assess primary care providers' contacts with study participants, including whether psychosocial concerns were identified since the injury.
Time Frame: 6 months
Reporting Status: Not Posted

7. Secondary Outcome: Health Service Utilization Over the 6 Months Post-injury
Description: Medical records were used as the primary source of service utilization data; parent report supplemented this information if records were unavailable.
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Intervention | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/39
Other Adverse Events (participants affected / at risk) | 0/46 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No